CLINICAL TRIAL: NCT00001756
Title: The Characterization of CD34+ Derived Mast Cell Precursors
Brief Title: Study of Mast Cell Precursors
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980027; 98-I-0027
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Mastocytosis; Healthy Volunteer
Keywords: Leukapheresis; Mastocytosis; Mast Cells; Normal Volunteer; Natural History; Systemic Mastocytosis
MeSH Terms: conditions — Mastocytosis; Mastocytosis, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood, Serum, White Cells

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy Volunteers
- Patients: Patients have mast cell hyperplasia compatible with a diagnosis of systemic mastocytosis (applicable to systemic mastocytosis patients only) or other allergic, hematologic, orimmunologic condition.

SUMMARY:
This study will investigate mast cell precursors that circulate in the blood. In a group of diseases collectively known as mastocytosis, mast cells accumulate in abnormal amounts in the skin, lymphoid tissues, bone marrow, liver and spleen. Some forms of mastocytosis have a generally good prognosis; for others, the prognosis is poorer. There is no known cure for any form of the disease. A better understanding of mast cells and how they respond to certain substances may provide insights that will lead to effective treatments for mastocytosis.

Patients with systemic mastocytosis and normal healthy volunteers between the ages of 20 and 60 may be eligible for this 8-day study. Participants will undergo the following procedures:

* Day 1 Medical history, physical examination, and blood tests to assess general health status
* Days 2 through 6 Daily injections under the skin of G-CSF a hormone that stimulates white blood cell production
* Day 7 Leukapheresis a procedure for collecting large numbers of white blood cells. In leukapheresis, blood is drawn through a needle placed in an arm and channeled into a cell separator machine. The white cells are collected and the rest of the blood is returned to the body through a needle in the other arm. The procedure takes up to 3 hours.
* Days 7 and 8 Blood draw (about 1 teaspoon) to monitor white blood cell counts.

DETAILED DESCRIPTION:
The purpose of this protocol is to obtain large numbers of CD34+ cells from the peripheral blood of healthy volunteers and patients with systemic mastocytosis or other related allergic, hematological, and immunological conditions by leukapheresis for culture and characterization of mast cell progenitor cells and their response to various cytokines and anti-mitotic agents. Healthy volunteers and patients will be adults of both sexes from 18 to 70 years of age. Granulocyte colony stimulating factor (G-CSF) will be administered to healthy volunteers at dose of 10 mcg/kg/day as a subcutaneous dose daily for 5 days not to exceed 960mcg. Patients will receive Plerixafor at a dose of 0.24 mg/kg as a single subcutaneous dose not to exceed 24mg the night before leukapheresis as a mobilizing agent for CD34+ cells. In identified patients where leukapheresis yield is considered adequate without stimulation by the principal investigator, leukapheresis may proceed without stimulation. Healthy volunteers will undergo a single leukapheresis at day 7, and patients will undergo a single leukapheresis at day 3 or 4. This is not a therapeutic protocol and does not involve reinfusion of any manipulated cells, viruses or DNA constructs back into human subjects.

ELIGIBILITY:
* SUBJECT INCLUSION CRITERIA:

Healthy Volunteers must:

1. Be 18-70 years of age
2. Be healthy
3. Have adequate peripheral venous access
4. Have normal renal function (creatinine less than or equal to 1.5mg/dL; less than or equal to 1 plus proteinuria)
5. Have normal hepatic function (bilirubin less than or equal to 1.5 mg/dL)
6. Have normal hematologic function (WBC greater than or equal to 3000/mm(3); granulocytes greater than or equal to 1500/mm(3) ; platelets greater than or equal to 175,000; hemoglobin greater than or equal to 12.5 g/dL)

Patients must:

1. Be 18-70 years of age
2. Have mast cell hyperplasia compatible with a diagnosis of systemic mastocytosis (applicable to systemic mastocytosis patients only) or other allergic, hematologic, or immunologic condition
3. Have adequate peripheral venous access or be willing to have a central line placed.
4. First be admitted as inpatients under an existing NIH protocol
5. Have preserved renal function (creatinine less than or equal to 2 mg/dL; less than or equal to 2 plus proteinuria)
6. Have preserved hepatic function (bilirubin less than or equal to 1.5 mg/dL)
7. Have preserved hematologic function (WBC greater than or equal to 3000/mm(3); granulocytes greater than or equal to 1500/mm(3) ; platelets greater than or equal to 175,000; hemoglobin greater than or equal to 12.5 g/dL)

All female subjects of childbearing potential:

1. May be enrolled if using effective contraception
2. Have a negative serum or urine pregnancy test determined within 72 hours before beginning Plerixafor or G-CSF administration

SUBJECT EXCLUSION CRITERIA:

All subjects must not meet any of the following criteria:

Healthy Volunteers and patients must not:

1. Have active bacterial, fungal or viral infections
2. Have viral screens positive for HIV or hepatitis B or C
3. Be pregnant or lactating
4. Have a history of autoimmune disease such as rheumatoid arthritis, vasculitis, pyoderma gangrenosum or similar disorder
5. Have any condition, which in the judgment of the investigator, might place the subject at undue risk

Healthy Volunteers with any of the following will be excluded:

1. Splenomegaly, pulmonary fibrosis and other related conditions
2. Use of any investigative drugs within the past 12 months
3. Have a significant coagulation disorder

Systemic Mastocytosis and Mast Cell Related Condition Patients with any of the following will be excluded:

1. Patients taking any other growth factors, cytokines or investigative drugs
2. Patients who are hemodynamically unstable (blood pressure systolic of lower than 105 or diastolic lower than 65)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Clinical
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 1997-12-03 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Use of G-CSF administration healthy volunteers to mobilize and enhance CD34+ hematopoietic progenitor cell numbers into the peripheral blood in order to culture and characterize human mast cells, study and characterize CD34+ -derived human ma... | 12/31/2029
  Use of G-CSF administration healthy volunteers to mobilize and enhance CD34+ hematopoietic progenitor cell numbers into the peripheral blood in order to culture and characterize human mast cells, study and characterize CD34+ -derived human mast cells.
Collection of CD34+ cells with or without use of Plerixafor administration in patients with systemic mastocytosis and other related allergic, hematological and immunological conditions to mobilize and enhance CD34+ cells into the peripheral b... | 12/31/2029
  Collection of CD34+ cells with or without use of Plerixafor administration in patients with systemic mastocytosis and other related allergic, hematological and immunological conditions to mobilize and enhance CD34+ cells into the peripheral blood to culture and learn how mast cells contribute to these disease states.

CONTACTS AND LOCATIONS:
Overall Officials: Melody C Carter, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Schwinger W, Mache C, Urban C, Beaufort F, Toglhofer W. Single dose of filgrastim (rhG-CSF) increases the number of hematopoietic progenitors in the peripheral blood of adult volunteers. Bone Marrow Transplant. 1993 Jun;11(6):489-92. PMID 8334430
- [Background] Metcalfe DD. Classification and diagnosis of mastocytosis: current status. J Invest Dermatol. 1991 Mar;96(3 Suppl):2S-4S; discussion 4S, 60S-65S. doi: 10.1111/1523-1747.ep12468882. PMID 16799601
- [Derived] Falduto GH, Pfeiffer A, Zhang Q, Yin Y, Metcalfe DD, Olivera A. A Critical Function for the Transcription Factors GLI1 and GLI2 in the Proliferation and Survival of Human Mast Cells. Front Immunol. 2022 Feb 16;13:841045. doi: 10.3389/fimmu.2022.841045. eCollection 2022. PMID 35251038
- [Derived] Wilson TM, Maric I, Simakova O, Bai Y, Chan EC, Olivares N, Carter M, Maric D, Robyn J, Metcalfe DD. Clonal analysis of NRAS activating mutations in KIT-D816V systemic mastocytosis. Haematologica. 2011 Mar;96(3):459-63. doi: 10.3324/haematol.2010.031690. Epub 2010 Dec 6. PMID 21134978
- [Derived] Prussin C, Lee J, Foster B. Eosinophilic gastrointestinal disease and peanut allergy are alternatively associated with IL-5+ and IL-5(-) T(H)2 responses. J Allergy Clin Immunol. 2009 Dec;124(6):1326-32.e6. doi: 10.1016/j.jaci.2009.09.048. PMID 20004787
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1998-I-0027.html